CLINICAL TRIAL: NCT03999970
Title: A Clinical Study to Develop a Sand Fly Biting Protocol Using Pathogen-free Blood-fed Sand Flies
Brief Title: A Clinical Study to Develop an Uninfected Sand Fly Biting Protocol
Acronym: FLYBITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of York (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Paul Kaye, Professor Paul Kaye, University of York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RE19_030_266151
Record Dates: First submitted 2019-05-23; First posted 2019-06-27 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Leishmaniasis, Cutaneous; Insect Bites
Keywords: Cutaneous Leishmaniasis; Controlled Human Infection Model; Sand Fly; Human Challenge
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Insect Bites and Stings

STUDY DESIGN:
Intervention Model Description: Clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phlebotomus papatasi sand fly bite (Active Comparator): Volunteers aged between 18-65 years will receive a bite or bites by sand flies using a watch-like biting chamber placed on the arm. The investigators will initially evaluate the use of biting chambers containing up to 5 sand flies maintained on the arm for 30 minutes, and evaluate the sand fly species Phlebotomus papatasi fed on blood twice in the laboratory prior to human exposure.
  Interventions: Other: Sand fly bite
- Phlebotomus duboscqi sand fly bite (Active Comparator): Volunteers aged between 18-65 years will receive a bite or bites by sand flies using a watch-like biting chamber placed on the arm. The investigators will initially evaluate the use of biting chambers containing up to 5 sand flies maintained on the arm for 30 minutes, and evaluate the sand fly species Phlebotomus duboscqi fed on blood twice in the laboratory prior to human exposure.
  Interventions: Other: Sand fly bite

INTERVENTIONS:
Other: Sand fly bite — Comparison between sand fly bites from two different species (Phlebotomus papatasi and Phlebotomus duboscqi)

SUMMARY:
The disease leishmaniasis mainly occurs in hot and tropical countries, affects millions of people and causes around 20,000 deaths across the world every year. Leishmaniasis is caused by the Leishmania parasite and is transmitted by sand flies. The parasite is tiny and not visible to the naked eye, whereas the particular sand fly is visible but small and inconspicuous. There are different types of leishmaniasis around the world and some can be very serious. They affect the skin (cutaneous leishmaniasis) or the internal organs of the body (visceral leishmaniasis). Some of the milder forms will produce skin problems which will be localised, whilst other forms of leishmaniasis will cause widespread skin changes. The skin lesions of cutaneous leishmaniasis can be disfiguring if left untreated.

There are some treatments for leishmaniasis available but many of them are not easy to use or don't work well. Therefore new treatments and vaccines are needed that prevent or work against leishmaniasis.

A solution being adopted for other diseases, which the investigators now wish to adopt for leishmaniasis is to develop a 'Controlled human infection model' (CHIM). These models involve deliberate exposure of individuals to an infection, in order to better understand how the disease works and to test potential vaccines and treatments. They have contributed vital scientific knowledge that has led to advances in the development of drugs and vaccines.

This is an initial study using uninfected (disease-free) sand flies, taking place at the University of York. The information from this study will help us to develop a model in the future using infected sand flies so that the investigators can assess any future vaccines against Leishmaniasis. The investigators will also hold a focus group after the sand fly biting study to explore the experiences of individuals taking part in this study.

DETAILED DESCRIPTION:
This is a healthy-volunteer clinical study to develop a sand fly biting protocol. 12 participants will be recruited for the study. It is an open-label randomized clinical study with 2 arms (for 2 different species of sand fly: Phlebotomus papatasi and Phlebotomus duboscqi). Participants will be randomized to each arm with 6 participants in each arm. This study will take place at the Translational Research Facility (Q Block), Hull York Medical School & Department of Biology, University of York, York.

The participants will be followed up to 21 days post-sand fly bite. There will then be a focus group once all participants have completed their follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 65 years on the day of screening
* Willing and able to give written informed consent
* Willing to undergo an Hepatitis B, Hepatitis C & HIV test
* Willing to undergo a pregnancy test during screening and follow-up visits and must not be breastfeeding (female volunteers)
* Willing to refrain from blood donation during the study
* Using a reliable and effective form of contraception (female volunteers)
* Judged, in the opinion of a medically qualified Clinical Investigator, to be able and likely to comply with all study requirements as set out in the protocol
* Without any other significant health problems as determined by medical history, physical examination, results of screening tests and the clinical judgment of a medically qualified Clinical Investigator
* Available for the duration of the study
* Willing to refrain from travel to regions where Leishmania-transmitting sand flies are present, from recruitment until the last study visit.
* Willing to consent to a report from the volunteer's GP (General Practitioner) confirming medical eligibility, to be provided before study entry

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

* Receipt of a live attenuated vaccine within 30 days or other vaccine within 14 days of screening
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned study.
* History of allergic disease/atopy or reactions or a history of severe or multiple allergies to drugs or pharmaceutical agents
* Any significant chronic skin condition as judged by the medical team
* Any history of Leishmaniasis
* Any history of travel within the last 30 days to regions where Leishmania major-transmitting sand flies are endemic*.
* Any past history of more than 30 contiguous days stay in regions where Leishmania major-transmitting sand flies are endemic*.
* Any history of severe local or general reaction to insect bites, defined as
* Local: extensive, indurated redness and swelling involving most of the antero-lateral thigh or the major circumference of the arm, not resolving within 72 hours
* General: fever ≥ 39.5°C within 48 hours, anaphylaxis, bronchospasm, laryngeal oedema, collapse, convulsions or encephalopathy within 48 hours
* Any history of anaphylaxis Females - pregnancy, less than 12 weeks postpartum, lactating or willingness/intention to become pregnant during the study and for 3 months following the study.
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Total IgE levels >81 Kilo-units/L Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months
* Tuberculosis, leprosy, or malnutrition
* Any chronic illness requiring hospital specialist input
* Any significant psychiatric conditions
* Any other significant disease, disorder or finding, which, in the opinion of a medically qualified Clinical Investigator, may either put the volunteer at risk because of participation in the study, or may influence the result of the study, or the volunteer's ability to participate in the study
* Unlikely to comply with the study protocol
* Involved in current or recent research within the past 3 months (as judged by study investigators) *This refers to regions where Leishmania major-transmitting sand flies are endemic including (but not limited to) the Middle East, Sub-Saharan Africa, and Asia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who successfully undergo sand fly bite during a 30 minute exposure determined by visual dermatoscopy | 21 days
  Development of a sand fly biting protocol using pathogen-free sand flies which is effective and safe for volunteers:
  Volunteers aged between 18-65 years will receive a bite or bites by sand flies using a watch-like biting chamber placed on the arm. The investigators will initially evaluate the use of biting chambers containing up to 5 sand flies maintained on the arm for 30 minutes, and evaluate the two sand fly species Phlebotomus papatasi and Phlebotomus duboscqi fed on blood twice in the laboratory prior to human exposure.

SECONDARY OUTCOMES:
Percentage of participants with visual changes following sand fly bite using photography. | 21 days
  The investigators will use photography to identify and record skin changes following sand fly bite by use of photography.
Percentage of participants with visual changes following sand fly bite using dermatoscopy. | 21 days
  The investigators will use dermatoscopy to identify and record skin changes following sand fly bite.
Percentage of participants with demonstrable serological evidence of sand fly bite. To determine human immunological response to sand fly bite using serology and cellular response measurement. | 21 days
  The investigators will measure serology including Leishmania and sand fly salivary gland antibodies following sand fly bite.
Percentage of participants with demonstrable cellular response evidence of sand fly bite. | 21 days
  The investigators will measure cellular response following sand fly bite
Percentage of participants with demonstrable evidence of change in IgE (immunoglobulin E) following sand fly bite. | 21 days
  The investigators will measure IgE at baseline and following sand fly bite
Percentage of participants with significant change in C-reactive protein following sand fly bite. | 21 days
  C-Reactive protein will be measured at baseline and following sand fly bite/
Determine size of lesion following sand fly bite over time | 21 days
  Rulers will be used to determine the changing size of any lesion

CONTACTS AND LOCATIONS:
Overall Officials: Charles Lacey, BMBS, MD, Principal Investigator — University of York
Locations (1):
- Translational Research Facility, Department of Biology, University of York, York, North Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Parkash V, Ashwin H, Sadlova J, Vojtkova B, Jones G, Martin N, Greensted E, Allgar V, Kamhawi S, Valenzuela JG, Layton AM, Jaffe CL, Volf P, Kaye PM, Lacey CJN. A clinical study to optimise a sand fly biting protocol for use in a controlled human infection model of cutaneous leishmaniasis (the FLYBITE study). Wellcome Open Res. 2021 Jun 30;6:168. doi: 10.12688/wellcomeopenres.16870.1. eCollection 2021. PMID 34693027
- [Derived] Parkash V, Jones G, Martin N, Steigmann M, Greensted E, Kaye P, Layton AM, Lacey CJ. Assessing public perception of a sand fly biting study on the pathway to a controlled human infection model for cutaneous leishmaniasis. Res Involv Engagem. 2021 May 30;7(1):33. doi: 10.1186/s40900-021-00277-y. PMID 34053461